CLINICAL TRIAL: NCT06172647
Title: Intestinal Microbiome Adherent to the Mucosa in Microscopic Colitis in Comparison With Patients With Advanced Colon Adenomas
Brief Title: Mucosa Adherent Intestinal Microbiome in Microscopic Colitis and Colorectal Cancer
Acronym: CMBACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Other Study IDs: P/22-066
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Microscopic Colitis; Colorectal Cancer; Colon Adenoma
Keywords: intestinal microbiome; mucosal adherent bacteria; dysbiosis; precancerous lesion
MeSH Terms: conditions — Colitis, Microscopic; Colorectal Neoplasms; Dysbiosis | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sigmoid tissue (colon)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Active Microscopic Colitis (MC) patients
  Interventions: Diagnostic Test: Colonoscopy
- Chronic watery diarrhoea patients
  Interventions: Diagnostic Test: Colonoscopy
- Patients with Advanced Colon Adenomas
  Interventions: Diagnostic Test: Colonoscopy
- Healthy controls
  Interventions: Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Endoscopic exploration of the colon (colonoscopy) for standard clinical practice (study of chronic watery diarrhoea, treatment of colon adenomas or population screening with a positive faecal occult blood test)

SUMMARY:
Microscopic colitis (MC) is an inflammatory bowel disease characterized by chronic non-bloody watery diarrhoea and a macroscopically normal colonic mucosa upon endoscopic exploration (colonoscopy). The diagnosis is performed by microscopic examination of mucosal biopsies that reveal specific histopathological change. Between 4-20% of patients with chronic non-bloody diarrhoea who undergo colonoscopy with serial biopsies are diagnosed with MC.

It has long been hypothesized that the microbiome plays a key role in the pathogenesis of MC. In patients with collagenous colitis, faecal stream diversion results in inflammation and histological remission, followed by disease relapse after intestinal transit is reconstructed. Moreover, studies carried out with faecal samples obtained after colonoscopy have demonstrated microbiome changes (reduced alpha diversity and higher microbial dysbiosis index) in patients with active MC. To avoid potential bias due to the effect of colonic lavage prior to colonoscopy in microbiota composition, the researchers of the present study previously evaluated the microbiome in faecal samples obtained before the diagnostic colonoscopy in patients with active MC. The results confirmed a reduced alpha diversity in diarrhoea groups; however, there were no differences between MC, bile-acid diarrhoea and functional diarrhoea. The microbial dysbiosis index was significantly higher in MC compared to the other diarrheal groups, but no bacterial species showed a significantly different relative abundance. On the other hand, the risk of colorectal cancer (CRC) or adenoma seems to be reduced in MC compared to controls. Growing evidence suggests microbial dysbiosis is a crucial environmental factor in the initiation of precancerous lesions of CRC such as adenomas.

The objective of the current multicentric prospective study is to assess the differences in the mucosa adherent intestinal microbiome between patients with MC, non-MC chronic diarrhoea, healthy controls and patients with advanced colon adenomas. In addition to the study of the microbiome, sociodemographic variables, history of drug usage, diets and specific characteristics of diarrhoea will be collected.

The hypothesis of the present study is that CM presents a specific mucosa adherent intestinal bacterial profile that may be relevant in the pathogenesis of the disease and that, additionally, may also play a protective role against the development of CRC and adenomas.

ELIGIBILITY:
Inclusion Criteria:

MC and Chronic watery diarrhea patients

1. Women ≥ 45 years old / Men ≥ 60 years old.
2. Patient with chronic watery diarrhea without blood with ≥2 liquid stools per day for minimum 3 times a week and lasting at least 1 month.
3. Blood analysis values within normality, with negative celiac disease serology and absence of acute phase reactants (normal C-reactive protein) and normal thyroid hormones. Calprotectin values may be elevated.
4. Signing of the informed consent.

Patients with Advanced Colon Adenomas

1. Age between 50 and 70 years.
2. Population screening participants with polyps with a crypt pattern of adenomatous appearance and polyp size of ≥10mm, or patients referred for endoscopic treatment of advanced adenomas.
3. Signing of the informed consent.

   Healthy controls

1. Age between 50 and 70 years. 2. Participants in the population screening with normal colonoscopy (without endoscopic alterations except presence of < 5 polyps (all less than 10mm) and/or colonic diverticulosis (except multiple diverticula in the sigma)). 3. Signing of the informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Patients who have received antibiotic, probiotic or prebiotic treatment in the 3 months prior to the study. 3. Patients who have traveled to developing or underdeveloped countries in the 3 months prior to the start of the study.

4. Patients who have received immunosuppressants and corticosteroids in the 3 months prior to the start of the study.

5. Patients who have received radiotherapy and/or chemotherapy in the 6 months prior to the start of the study.

6. Consumption of herbal products. 7. Bacterial or parasitic intestinal infection (including Blastocystis hominis).

8. History of inflammatory bowel disease or celiac disease. 9. Previous gastrointestinal surgery (excluding appendectomy or inguinal hernia repair).

10. Incomplete colonoscopy or lack of biopsies of the right, transverse and left colon.

11. Unsatisfactory preparation for a complete examination (Boston scale <6, any segment <2).

12. Inability to understand the instructions involved in participating in this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from participating centers that require a colonoscopy for standard clinical practice (study of chronic watery diarrhoea, treatment of colon adenomas or population screening with a positive faecal occult blood test)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion and abundance of bacterial taxa (defined as total percentage of bacterial DNA sequences) | at inclusion (colonoscopy)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari MútuaTerrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Background] Miehlke S, Guagnozzi D, Zabana Y, Tontini GE, Kanstrup Fiehn AM, Wildt S, Bohr J, Bonderup O, Bouma G, D'Amato M, Heiberg Engel PJ, Fernandez-Banares F, Macaigne G, Hjortswang H, Hultgren-Hornquist E, Koulaouzidis A, Kupcinskas J, Landolfi S, Latella G, Lucendo A, Lyutakov I, Madisch A, Magro F, Marlicz W, Mihaly E, Munck LK, Ostvik AE, Patai AV, Penchev P, Skonieczna-Zydecka K, Verhaegh B, Munch A. European guidelines on microscopic colitis: United European Gastroenterology and European Microscopic Colitis Group statements and recommendations. United European Gastroenterol J. 2021 Feb 22;9(1):13-37. doi: 10.1177/2050640620951905. Online ahead of print. PMID 33619914
- [Background] Jarnerot G, Tysk C, Bohr J, Eriksson S. Collagenous colitis and fecal stream diversion. Gastroenterology. 1995 Aug;109(2):449-55. doi: 10.1016/0016-5085(95)90332-1. PMID 7615194
- [Background] Rindom Krogsgaard L, Kristian Munck L, Bytzer P, Wildt S. An altered composition of the microbiome in microscopic colitis is driven towards the composition in healthy controls by treatment with budesonide. Scand J Gastroenterol. 2019 Apr;54(4):446-452. doi: 10.1080/00365521.2019.1599064. Epub 2019 Apr 22. PMID 31009268
- [Background] Morgan DM, Cao Y, Miller K, McGoldrick J, Bellavance D, Chin SM, Halvorsen S, Maxner B, Richter JM, Sassi S, Burke KE, Yarze JC, Ludvigsson JF, Staller K, Chung DC, Khalili H. Microscopic Colitis Is Characterized by Intestinal Dysbiosis. Clin Gastroenterol Hepatol. 2020 Apr;18(4):984-986. doi: 10.1016/j.cgh.2019.06.035. Epub 2019 Jun 27. PMID 31254673
- [Background] Shobar RM, Velineni S, Keshavarzian A, Swanson G, DeMeo MT, Melson JE, Losurdo J, Engen PA, Sun Y, Koenig L, Mutlu EA. The Effects of Bowel Preparation on Microbiota-Related Metrics Differ in Health and in Inflammatory Bowel Disease and for the Mucosal and Luminal Microbiota Compartments. Clin Transl Gastroenterol. 2016 Feb 11;7(2):e143. doi: 10.1038/ctg.2015.54. PMID 26866392
- [Background] Drago L, Valentina C, Fabio P. Gut microbiota, dysbiosis and colon lavage. Dig Liver Dis. 2019 Sep;51(9):1209-1213. doi: 10.1016/j.dld.2019.06.012. Epub 2019 Jul 27. PMID 31358483
- [Background] Batista L, Robles V, Manichanh C, Ruiz L, Guagnozzi D, Pinsach F, Guarner F, Fernandez-Banares F. Colonic bacterial diversity and dysbiosis in active microscopic colitis as compared to chronic diarrhoea and healthy controls: effect of polyethylene glycol after bowel lavage for colonoscopy. BMC Gastroenterol. 2022 Jun 28;22(1):320. doi: 10.1186/s12876-022-02392-w. PMID 35764931
- [Background] Aprile F, Bruno G, Palma R, Mascellino MT, Panetta C, Scalese G, Oliva A, Severi C, Pontone S. Microbiota Alterations in Precancerous Colon Lesions: A Systematic Review. Cancers (Basel). 2021 Jun 19;13(12):3061. doi: 10.3390/cancers13123061. PMID 34205378